CLINICAL TRIAL: NCT00516750
Title: Phase II Clinical Trial Concerning Gene Expression Profiling to Predict the Chemosensitivity of Invasive Bladder Cancer
Brief Title: Gene Expression Profiling in Patients With Invasive Bladder Cancer Receiving Methotrexate, Vinblastine, Doxorubicin, and Cisplatin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of enrollment.
Sponsor: Kyoto University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: TRIC-UHA-GU-03-01; CDR0000561303 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2008-03

CONDITIONS: Bladder Cancer
Keywords: recurrent bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Doxorubicin; Methotrexate; Vinblastine; Gene Expression Profiling; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: methotrexate
Drug: vinblastine
Genetic: gene expression profiling
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methotrexate, vinblastine, doxorubicin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Evaluating blood or tissue samples from patients with cancer may help doctors learn more about changes that occur in DNA, identify biomarkers related to cancer, and predict how well patients will respond to combination chemotherapy.

PURPOSE: This phase II trial is studying gene expression profiling to see how well it works in predicting response to treatment in patients with invasive bladder cancer receiving methotrexate, vinblastine, doxorubicin, and cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Analyze the correlation between gene expression profile and the effect of chemotherapy and detect the significant cluster of genes useful to predict chemosensitivity.
* Confirm the reduction in original tumor size in patients with invasive bladder cancer treated with methotrexate, vinblastine, doxorubicin hydrochloride, and cisplatin.

Secondary

* Determine the safety of this regimen in these patients.
* Determine the overall survival rate in patients treated with this regimen.
* Assess the reduction in size of metastatic lesions in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive methotrexate on days 1, 15, and 22, vinblastine on days 2, 15, and 22, doxorubicin hydrochloride and cisplatin on day 2. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patient samples will be collected for gene expression profiling.

After completion of study treatment, patients are followed for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of invasive bladder cancer
* Must be confirmed by chest and abdominal CT scan OR pelvic MRI scan and transurethral biopsy (with definitive muscle invasion > T2) within 4 weeks prior to registration

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,000/mm^3
* Neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 mg/dL
* Serum creatinine ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 x upper limit of normal
* Not pregnant
* No liver cirrhosis
* No ischemic cardiovascular disease or arrhythmia for which treatment is necessary
* No cardiac infarction within the past 6 months
* No interstitial pneumonia, pulmonary fibrosis, or any other diseases by which oxygen inhalation therapy is needed
* No active cancerous lesion other than upper urinary tract tumor
* No high fever or any other infectious symptom
* No uncontrolled hypertension or diabetes mellitus

PRIOR CONCURRENT THERAPY:

* No prior systemic chemotherapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Detection of genes associated with sensitivity to the chemotherapy in tumor size reduction of original bladder tumor

SECONDARY OUTCOMES:
Safety
Overall survival rate
Size reduction of metastatic lesion

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ogawa, MD, PhD, Study Chair — Kyoto University Hospital
Locations (5):
- Japan (5):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kyoto University Hospital, Kyoto, Kyoto
  - National Hospital Organization - Kyoto Medical Center, Kyoto, Kyoto
  - Shiga Medical Center for Adults, Moriyama, Shiga
  - Osaka Red Cross Hospital, Osaka